CLINICAL TRIAL: NCT01875198
Title: Oncologic Impact of Splenectomy-omitting Radical Pancreatectomy in Well-selected Left-sided Pancreatic Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: because of difficulties of enrolling appropriate participants
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0138
Record Dates: First submitted 2013-05-28; First posted 2013-06-11 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Left-sided Pancreatic Cancer; Ductal Adenocarcinoma
Keywords: Splenectomy;; Spleen-preserving
MeSH Terms: interventions — Splenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RAMPS (Experimental): Radical Antegrade Modular Pancreatectomy with Splenectomy
  Interventions: Procedure: Radical Antegrade Modular Pancreatectomy with Splenectomy
- RAMP (Active Comparator): Radical Antegrade Modular Pancreatectomy without splenectomy
  Interventions: Procedure: Radical Antegrade Modular Pancreatectomy without splenectomy

INTERVENTIONS:
Procedure: Radical Antegrade Modular Pancreatectomy with Splenectomy
  Arms: RAMPS
Procedure: Radical Antegrade Modular Pancreatectomy without splenectomy — distal pancreatectomy without pancreatectomy
  Arms: RAMP

SUMMARY:
When distal pancreatectomy is carried out for left-sided pancreatic cancer, splenectomy is usually performed not only for margin-negative resection but also for effective clearance of the splenic hilar lymph nodes. However, there was no scientific evidence regarding the justifiability for spleen resection. Considering potential immunological function of the spleen, the investigators hypothesized that distal pancreatectomy without pancreatectomy for left-sided pancreatic cancer is superior than Distal pancreatectomy with pancreatectomy in terms of short-term perioperative outcomes and disease-specific overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Ductal adenocarcinoma
2. Age ≥20 and ≤80
3. General performance status: the Karnofsky score> 70% or ECOG 0-1
4. Potentially Curative resection
5. Tumor size < 3cm
6. Pancreatic cancer located on neck or body portion
7. No invasion to spleen or spleen hilum
8. No combined resection except Lt. adrenal gland
9. Distance more than 5cm (≥5cm) between tumor lateral margin and spleen hilum

Exclusion Criteria:

1. Unresectable or locally advanced, metastatic case
2. Patients who do not want surgery
3. ASA (American society of anesthesiologists' physical status classification) score: ≥3
4. Patients with drug or alcohol addiction
5. Patients showing low compliance
6. Patients who not want to involve the clinical trial
7. Patients who are unable to read or understand the informed consent, sign a consent form (eg, mental retardation, blindness, illiteracy, foreign, etc.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Bleeding amount | 5 hours

SECONDARY OUTCOMES:
average of pain score | admission period(about 5 days)
time interval to adjuvant treatment | admission period(about 5 days)
postoperative complication | admission period(about 5 days)
  (e.g. postoperative pancreatic fistula, delayed gastric emptying, intra-abdominal abscess, postoperative bleeding, wound infection, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Kim SH, Kang CM, Satoi S, Sho M, Nakamura Y, Lee WJ. Proposal for splenectomy-omitting radical distal pancreatectomy in well-selected left-sided pancreatic cancer: multicenter survey study. J Hepatobiliary Pancreat Sci. 2013 Mar;20(3):375-81. doi: 10.1007/s00534-012-0549-z. PMID 22911134